CLINICAL TRIAL: NCT04505839
Title: First-In-Human Dose-Escalation Study of STP1002 in Patients With Advanced-Stage Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ST Pharm Co., Ltd. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP-ST-01
Record Dates: First submitted 2020-08-02; First posted 2020-08-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STP1002 (Experimental)
  Interventions: Drug: STP1002

INTERVENTIONS:
Drug: STP1002 — Oral capsule, QD
  Other Names: Basroparib

SUMMARY:
This is an open-label, multicenter, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics (PK) and to determine the maximum tolerated dose (MTD) of STP1002 in patients with advanced-stage solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced-stage solid tumor (metastatic or locally advanced and unresectable) with histologically confirmed diagnosis of CRC, NSCLC, GC, RCC, or HCC
* Measurable lesion(s) according to RECIST 1.1 criteria
* Performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Ability to swallow capsules
* Received last chemotherapy, biologic, or investigational therapy at least 4 weeks prior to first dosing of study treatment
* Has received or is intolerant to all standard of care treatment options with known clinical benefit
* Life expectancy of more than 3 months
* Adequate hematological, hepatic and renal function
* For women of childbearing potential, a negative serum pregnancy test performed within 7 days prior to start of treatment

Exclusion Criteria:

* Received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Major surgery within the last 28 days prior to the first dose of investigational drug
* Prior radiation therapy within 14 days prior to study Cycle 1 Day 1 and/or persistence of radiation-related adverse effects.
* Concurrent treatment with any anticancer agent
* Currently taking either strong CYP inhibitors or inducers
* Known brain metastases, uncontrolled seizure disorder, or active neurologic disease
* Significant cardiovascular impairment
* Pregnant or nursing
* Known HIV infection, active hepatitis C and/or hepatitis B infection
* Known bleeding disorder or coagulopathy
* Active drug or alcohol abuse or history of alcohol or drug abuse during the last two years.
* Diagnosis of osteoporosis at the time of the screening
* Any history of retinal pathology including diabetic retinopathy, macular degeneration, or other retinal degenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 28 days
  DLTs are defined as any of the following adverse events (AEs) that are possibly or probably related to the trial regimen occurring during Cycle 1

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | 24 months
  Number and severity of TEAEs, treatment-related AEs, and SAEs for all dose groups according to the NCI CTCAE v5.0
The pharmacokinetics of STP1002 | 24 months
  Plasma concentration of STP1002 following oral administration

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Northwestern University, Evanston, Illinois